CLINICAL TRIAL: NCT00848042
Title: A Pilot Study of AuroLase(tm) Therapy in Patients With Refractory and/or Recurrent Tumors of the Head and Neck
Brief Title: Pilot Study of AuroLase(tm) Therapy in Refractory and/or Recurrent Tumors of the Head and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanospectra Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-07-001
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Cancer
Keywords: cancer; head and neck; laser; ablation
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AuroShell-3.5 (Active Comparator): Group treated with the lowest treatment level with 4.5 ml/Kg of AuroShell particles concentrated to 100 optical density and 3.5 watts. Device: AuroLase Therapy
  Interventions: Device: AuroLase Therapy
- AuroShell-4.5 (Active Comparator): Group treated with up to 7.5 ml/Kg of AuroShell particles concentrated to 100 optical density and 4.5 watts. Device: AuroLase Therapy
  Interventions: Device: AuroLase Therapy
- AuroShell-5.0 (Active Comparator): Group treated with up to 7.5 ml/Kg of AuroShell particles concentrated to 100 optical density and 5.0 watts. Device: AuroLase Therapy
  Interventions: Device: AuroLase Therapy

INTERVENTIONS:
Device: AuroLase Therapy — Infusion of AuroShell particles followed by laser illumination for photothermal ablation of target lesions

SUMMARY:
This is an open-label, multicenter, single-dose pilot study of AuroLase(TM) Therapy in the treatment of patients with refractory and/or recurrent tumors of the head and neck. Three (3) treatment groups of five (5) patients each will be enrolled and observed for six (6) months following treatment. Each group will receive a single dose of AuroShell(TM) particles followed by one or more interstitial illuminations with an 808nm laser. Particle dose and laser power may be increased in each dosing group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented histological or cytological evidence of tumor(s) of the head and neck
* Patients must have one or more refractory and/or recurrent tumors of the head and neck which have at least one dimension with longest diameter 15 mm using conventional techniques or 10 mm with spiral CT scan.
* Target lesions should be accessible to examination (examination by fiber optic nasopharyngoscopy or laryngoscopy is permitted) and to biopsy.
* Each index lesion should be large enough to provide at least 6 mg of tumor tissue by biopsy (such as an 18 gauge Tru-Cut needle biopsy 1cm in length or similar technique) for assessment by neutron activation analysis.
* Tumors must be measurable according to RECIST criteria
* Patients must be ≥ 18 years of age
* Patients must have ECOG Performance Score of 0, 1 or 2 (see Appendix 3)
* Patients or their legal representative must be able to read, understand and sign an informed consent
* Adequate renal function as evidenced by serum creatinine ≤ 2.0 mg/dL
* Adequate hepatic function as evidenced by: Serum total bilirubin ≤ 2.0 mg/dL, Alkaline phosphatase ≤ 2X the ULN for the reference lab, SGOT/SGPT ≤ 2X the ULN for the reference lab
* Women of childbearing potential must agree to use an effective form of contraception during the study and for 90 days following treatment (an effective form of contraception is an oral contraceptive or a double barrier method). Women who are NOT of childbearing potential are those who have undergone a bilateral oophorectomy or who have undergone menopause, defined as an absence of a menstrual cycle for 12 consecutive months.
* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Patients with known hypersensitivity to any of the components of the PEGylated AuroShell suspension (polyethylene glycol, gold)
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within a period of 5 half-lives of the investigational therapy in question prior to the day of dosing with the PEGylated AuroShell particles (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Patients who are pregnant and/or lactating
* Patients with evidence of an active bacterial infection or with a fever ≥ 38.5 ºC (101.3 ºF) within 3 days of the first scheduled day of dosing
* Patients who have undergone splenectomy
* Patient who has had a course of radiotherapy in the treatment area within the past 30 days.
* Patient who has had a course of chemotherapy or other anti-neoplastic therapy in the past 30 days.
* Patient who has had surgery within 2 cm of the treatment area within the past two weeks.
* Life expectancy of less than 3 months.
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cancer Treatment Centers of American Western Regional Medical Center, Goodyear, Arizona
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects screened and enrolled at four sites in the United States.
Groups:
- AuroShell-3.5: Group treated with the lowest treatment level with 4.5 ml/Kg of AuroShell particles concentrated to 100 Optical Density and 3.5 watts.
- AuroShell-4.5: Group treated with up to 7.5 ml/Kg of AuroShell particles concentrated to 100 Optical Density and 4.5 watts.
- AuroShell-5.0: Group treated with up to 7.5 ml/Kg of AuroShell particles concentrated to 100 Optical Density and 5 watts.
Period: Overall Study
Arm/Group | AuroShell-3.5 | AuroShell-4.5 | AuroShell-5.0
Started | 5 | 5 | 1
Day 1 | 5 | 5 | 1
Day 2 | 5 | 5 | 1
Day 3 | 5 | 5 | 1
Day 8 | 5 | 5 | 1
Day 15 | 4 | 5 | 1
Month 1 | 4 | 5 | 1
Month 2 | 1 | 5 | 1
Month 3 | 1 | 4 | 1
Month 4 | 1 | 4 | 1
Month 5 | 1 | 3 | 1
Month 6 | 1 | 3 | 1
Completed | 1 | 3 | 1
Not Completed | 4 | 2 | 0
Not completed — Death | 1 | 2 | 0
Not completed — Other Therapy | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AuroShell-3.5 | AuroShell-4.5 | AuroShell-5.0 | Total
Number analyzed (Participants) | 5 | 5 | 1 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 1 | 7
  >=65 years | 2 | 2 | 0 | 4
Gender [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 4 | 4 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 3 | 5 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 5 | 4 | 0 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Device Effects Considered Attributable to AuroShell Particle Administration
Description: Includes all participants that experienced an adverse device effect that were rated probable or definitely related to AuroShell particle infusion
Time Frame: up to 6 months
Population: per protocol
Measure: Number; unit: participants
Arm/Group | AuroShell-3.5 | AuroShell-4.5 | AuroShell-5.0
Number analyzed (Participants) | 5 | 5 | 1
participants | 2 | 2 | 0

2. Secondary Outcome: Response in Targeted Tumors.
Time Frame: 6 months
Population: Data was not collected/analyzed
Arm/Group | AuroShell-3.5 | AuroShell-4.5 | AuroShell-5.0
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months post-study
Description: If a subject experienced more than one event, the subject is only counted once for the most severe event. If a subject experience more than one event in an system class, the subject is only counted once.
  All adverse events are being reported regardless of relation to study treatment.
Arm/Group | AuroShell-3.5 | AuroShell-4.5 | AuroShell-5.0
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/5 | 0/1
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AuroShell-3.5 (N=5) | AuroShell-4.5 (N=5) | AuroShell-5.0 (N=1)
Cardiac Event (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasm, Mouth (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Numbness (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AuroShell-3.5 (N=5) | AuroShell-4.5 (N=5) | AuroShell-5.0 (N=1)
Anemia, Unspecified (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis, Unspecified (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema, NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal Reflux (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension, Unspecified (General disorders) | 2 (2) | 1 (1) | 0 (0)
Sinus Tachycardia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain, Neoplasm Related (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Pytalism (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other